CLINICAL TRIAL: NCT00571896
Title: The Use of SennaS for Prevention of Post-operative Constipation After Urogynecologic Surgery: a Randomized Double Blinded Placebo Controlled Trial
Brief Title: The Use of SennaS for Prevention of Post-operative Constipation After Urogynecologic Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PATE002472HE
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Constipation
Keywords: constipation; SennaS
MeSH Terms: conditions — Constipation | interventions — doxidan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SennaS (Experimental): This group of participants will receive SennaS to use after surgery.
  Interventions: Drug: Senna+ docusate
- Placebo (Placebo Comparator): This group of participants will receive placebo pills to use after surgery.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Senna+ docusate — Senna+Docusate: dose will be 8.6 mg senna concentrate with 50 mg docusate. The participants will take the medication as follows: 1. Drink 4-6 glasses of fluid a day for the first two weeks after surgery 2. Take 2 SennaS tabs at bedtime the first night home from the hospital 3. If no bowel movement that next morning, take 2 tabs after breakfast. 4. If no bowel movement by evening, take 3 tabs at bedtime 5. If no bowel movement that next morning, take 3 tabs after breakfast 6. Once you do have a bowel movement, use the regimen described in the step two steps prior to the last one you used as your daily regimen. So, if you had a BM the morning after 3 tabs at bedtime, use steps 2 & 3 (2 tabs at night and in the morning) until the first-postoperative visit.
  Other Names: SennaS or Senokot-S
  Arms: SennaS
Drug: placebo — Placebo pill: The participants will use the placebo pills in the following manner: 1. Drink 4-6 glasses of fluid a day for the first two weeks after surgery 2. Take 2 SennaS tabs at bedtime the first night home from the hospital 3. If no bowel movement that next morning, take 2 tabs after breakfast. 4. If no bowel movement by evening, take 3 tabs at bedtime 5. If no bowel movement that next morning, take 3 tabs after breakfast 6. Once you do have a bowel movement, use the regimen described in the step two steps prior to the last one you used as your daily regimen. So, if you had a BM the morning after 3 tabs at bedtime, use steps 2 & 3 (2 tabs at night and in the morning) until the first-postoperative visit.
  Other Names: Blank pill
  Arms: Placebo

SUMMARY:
We are doing this study to see if using an over the counter mild laxative, SennaS, there is a difference in time required to have a bowel movement in women who are having surgery for prolapse (when your uterus and/or vagina drop after childbirth or with age) and/or incontinence (when you leak urine or stool without your control) as compared to a sugar pill or placebo.

DETAILED DESCRIPTION:
Right now, doctors use mild laxatives and stool softeners to help you have a bowel movement earlier and with less pain after surgery. Sometimes if the stool softener or mild laxatives do not work, you may need to use stronger laxatives or enemas. We want to see if specifically using SennaS is better for having a bowel movement soon after surgery and with less pain. SennaS is FDA approved for constipation. It has a stool softener and a mild laxative and has been shown to be safe and effective for treating constipation.

ELIGIBILITY:
Inclusion Criteria:

Women undergoing pelvic reconstructive surgery, including any combination of:

* Posterior/rectocele repair
* Paravaginal repair
* Anterior/cystocele repair
* Suburethral sling
* Abdominal sacrocolpopexy
* Midurethral sling (obturator pass)
* Burch urethropexy
* Midurethral sling (retropubic pass)
* Colpocleisis/colpectomy
* Uterosacral ligament suspension
* Sacrospinous ligament fixation
* Enterocele repair
* Anal sphincter repair
* Perineorrhaphy
* Use of graft material (synthetic or biologic) of any form/size does not affect inclusion, use of laparoscopy or robotic-assisted laparoscopy does not affect inclusion

Exclusion Criteria:

* Male
* Pregnancy (based on positive urine or serum ß-HCG measurement preoperatively in women who are not menopausal or have prior hysterectomy)
* Concurrent bowel resection,
* Hirschsprung's Disease or gastroparesis,
* Irritable & inflammatory bowel disease (Crohn's Disease/ulcerative colitis) formally diagnosed,
* Clostridium difficile colitis during present hospitalization
* Inability to understand written study material,
* Inability to give consent
* Rectal bleeding or presently diagnosed colorectal cancer,
* Documented preoperative daily use of SennaS for more than 3 weeks,
* Known allergy to SennaS
* Inability to use suppositories/enemas

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
1. Time to first bowel movement after surgery. 2. Need for magnesium citrate or enemas in the immediate post-operative period. | 7 weeks post-operatively

SECONDARY OUTCOMES:
Straining and pain with bowel movements in the immediate post-operative period | First post-operative week

CONTACTS AND LOCATIONS:
Overall Officials: Christine A LaSala, MD, Principal Investigator — Hartford Hospital, Division of Urogynecology
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

REFERENCES:
- [Background] Jewell DJ, Young G. Interventions for treating constipation in pregnancy. Cochrane Database Syst Rev. 2001;(2):CD001142. doi: 10.1002/14651858.CD001142. PMID 11405974
- [Background] Kochen MM, Wegscheider K, Abholz HH. Prophylaxis of constipation by wheat bran: a randomized study in hospitalized patients. Digestion. 1985;31(4):220-4. doi: 10.1159/000199203. PMID 2989052
- [Background] Schmelzer M. Effectiveness of wheat bran in preventing constipation of hospitalized orthopaedic surgery patients. Orthop Nurs. 1990 Nov-Dec;9(6):55-9. doi: 10.1097/00006416-199011000-00010. PMID 2177180
- [Background] Kacmaz Z, Kasici M. Effectiveness of bran supplement in older orthopaedic patients with constipation. J Clin Nurs. 2007 May;16(5):928-36. doi: 10.1111/j.1365-2702.2006.01766.x. PMID 17462043
- [Background] Franneby U, Gunnarsson U, Wollert S, Sandblom G. Discordance between the patient's and surgeon's perception of complications following hernia surgery. Hernia. 2005 May;9(2):145-9. doi: 10.1007/s10029-004-0310-x. Epub 2005 Feb 10. PMID 15703861
- [Background] Corman ML. Management of postoperative constipation in anorectal surgery. Dis Colon Rectum. 1979 Apr;22(3):149-51. doi: 10.1007/BF02586804. PMID 87299
- [Background] Jelovsek JE, Barber MD, Paraiso MF, Walters MD. Functional bowel and anorectal disorders in patients with pelvic organ prolapse and incontinence. Am J Obstet Gynecol. 2005 Dec;193(6):2105-11. doi: 10.1016/j.ajog.2005.07.016. PMID 16325624
- [Background] Arya LA, Novi JM, Shaunik A, Morgan MA, Bradley CS. Pelvic organ prolapse, constipation, and dietary fiber intake in women: a case-control study. Am J Obstet Gynecol. 2005 May;192(5):1687-91. doi: 10.1016/j.ajog.2004.11.032. PMID 15902178
- [Background] Bradley CS, Brown MB, Cundiff GW, Goode PS, Kenton KS, Nygaard IE, Whitehead WE, Wren PA, Weber AM; Pelvic Floor Disorders Network. Bowel symptoms in women planning surgery for pelvic organ prolapse. Am J Obstet Gynecol. 2006 Dec;195(6):1814-9. doi: 10.1016/j.ajog.2006.07.008. Epub 2006 Sep 25. PMID 16996465
- [Background] da Silva GM, Gurland B, Sleemi A, Levy G. Posterior vaginal wall prolapse does not correlate with fecal symptoms or objective measures of anorectal function. Am J Obstet Gynecol. 2006 Dec;195(6):1742-7. doi: 10.1016/j.ajog.2006.07.034. PMID 17132476
- [Background] Lewis SJ, Heaton KW. Stool form scale as a useful guide to intestinal transit time. Scand J Gastroenterol. 1997 Sep;32(9):920-4. doi: 10.3109/00365529709011203. PMID 9299672
- [Background] Mahony R, Behan M, O'Herlihy C, O'Connell PR. Randomized, clinical trial of bowel confinement vs. laxative use after primary repair of a third-degree obstetric anal sphincter tear. Dis Colon Rectum. 2004 Jan;47(1):12-7. doi: 10.1007/s10350-003-0009-6. Epub 2004 Jan 14. PMID 14719145
- [Background] Griffenberg L, Morris M, Atkinson N, Levenback C. The effect of dietary fiber on bowel function following radical hysterectomy: a randomized trial. Gynecol Oncol. 1997 Sep;66(3):417-24. doi: 10.1006/gyno.1997.4797. PMID 9299255
- [Background] Frank L, Kleinman L, Farup C, Taylor L, Miner P Jr. Psychometric validation of a constipation symptom assessment questionnaire. Scand J Gastroenterol. 1999 Sep;34(9):870-7. doi: 10.1080/003655299750025327. PMID 10522604